CLINICAL TRIAL: NCT00440648
Title: A Double-Blind, Cross-Over Design Study of Sevelamer Hydrochloride (Renagel®) and Sevelamer Carbonate in Chronic Kidney Disease Patients on Hemodialysis
Brief Title: Cross-Over Study of Sevelamer Hydrochloride and Sevelamer Carbonate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GD3-163-201
Record Dates: First submitted 2007-02-24; First posted 2007-02-27 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Other): sevelamer carbonate w(1-8) sevelamer hydrochloride w(9-16)
  Interventions: Drug: sevelamer carbonate, sevelamer hydrochloride
- 2 (Other): sevelamer hydrochloride w(1-8) sevelamer carbonate w(9-16)
  Interventions: Drug: sevelamer hydrochloride, sevelamer carbonate

INTERVENTIONS:
Drug: sevelamer carbonate, sevelamer hydrochloride — Starting dose individualized for each patient and fixed daily dose throughout both treatment periods
  Arms: 1
Drug: sevelamer hydrochloride, sevelamer carbonate — Starting dose individualized for each patient and fixed daily dose throughout both treatment periods
  Arms: 2

SUMMARY:
This is a double-blind, randomized, cross-over study conducted at centers within the United States. The study consists of five periods: an up to two-week Screening Period, a 5-week Run-In Period, two eight-week study treatment periods and a two-week Washout Period. Patients are assigned randomly (1:1) to one of two treatment sequences: sevelamer carbonate for eight weeks followed by sevelamer hydrochloride for eight weeks or sevelamer hydrochloride for eight weeks followed by sevelamer carbonate for eight weeks

DETAILED DESCRIPTION:
The study was conducted at 15 centers (2 of which did not enroll any patients). A total of 79 hemodialysis patients were assigned randomly to one of two treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

* patient had received hemodialysis three times per week for 3 months or longer;
* patients were maintained on sevelamer hydrochloride as their primary phosphate binder with a total daily dose of ≤ 13.6 g with serum phosphorus concentrations at the last two measurements between 3.0 and 6.5 mg/dL, the most recent iPTH ≤ 600 pg/mL and the most recent serum calcium within the normal range.

Exclusion Criteria:

* if patient had active bowel obstruction, dysphagia, swallowing disorders, or severe gastrointestinal motility disorders;
* active ethanol or drug abuse (excluding tobacco);
* need for antidysrhythmic or antiseizure medications used to control these conditions;
* poorly controlled diabetes mellitus or hypertension;
* active vasculitis;
* active malignancy other than basal-cell carcinoma;
* HIV infection; or
* any clinically significant unstable medical condition as judge by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety-evaluated on the basis of adverse events (reported and/or observed) | 16 weeks
changes in laboratory parameters, vital signs | 16 weeks
note: clinically significant changes in physical examination were recorded and evaluated as adverse events | 16 weeks
Efficacy-treatment regimens are compared on the basis of serum phosphorus at the end of each treatment period using the time-weighted mean of the phosphorus value from the last three visits in each treatment period | 16 weeks
Treatment regimens were also compared with respect to total, LDL, and HDL cholesterol, and triglycerides, using the mean of values for each parameter from the two post-baseline assessments in each treatment period. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (14):
- United States (14):
  - Mobile, Alabama
  - Riverside, California
  - Greenwood Village, Colorado
  - Berwyn, Illinois
  - Crestwood, Illinois
  - Indianapolis, Indiana
  - Valparaiso, Indiana
  - Columbus, Missouri
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Easton, Pennsylvania
  - Wynnewood, Pennsylvania
  - Nashville, Tennessee
  - Norfolk, Virginia